CLINICAL TRIAL: NCT02937298
Title: The Thermic Effect of Some Plant Foods Native to Scotland: A Pilot Study.
Brief Title: Thermic Effects of Some Scottish Plant Foods
Acronym: ThermicFoods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016/RINH/2
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Diet Induced Thermogenesis; Obesity Control
Keywords: Diet Induced Thermogenesis; Obesity; Energy balance; Energy expenditure; berries; Sea Buckthorn; Wild garlic
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control Meal (Experimental): Control meal using standard breakfast foods.
  Interventions: Dietary Supplement: Control Meal
- Berry Treatment (Experimental): This will consist of standard breakfast foods plus a berry smoothie.
  Interventions: Dietary Supplement: Berry Treatment
- Sea Buckthorn Treatment (Experimental): This will consist of standard breakfast foods plus a sea buckthorn berry smoothie.
  Interventions: Dietary Supplement: Sea Buckthorn Treatment
- Wild Garlic Treatment (Experimental): This will consist of standard breakfast foods plus a wild garlic dip.
  Interventions: Dietary Supplement: Wild Garlic Treatment

INTERVENTIONS:
Dietary Supplement: Control Meal — This will consist of standard breakfast foods (cereal, milk, yoghurt, cheese cracker bread, butter, banana and cream
  Arms: Control Meal
Dietary Supplement: Berry Treatment — This will consist of standard breakfast foods (cereal, milk, yoghurt, cheese cracker bread, butter, banana and cream plus a berry smoothie. The berry smoothie consists of blueberries, raspberries and blackberries.
  Arms: Berry Treatment
Dietary Supplement: Sea Buckthorn Treatment — This will consist of standard breakfast foods (cereal, milk, yoghurt, cheese cracker bread, butter, banana and cream plus a sea buckthorn berry smoothie.
  Arms: Sea Buckthorn Treatment
Dietary Supplement: Wild Garlic Treatment — This will consist of standard breakfast foods (cereal, milk, yoghurt, cheese cracker bread, butter, banana and cream. The wild garlic will be prepared and served as a dip alongside.
  Arms: Wild Garlic Treatment

SUMMARY:
Weight gain occurs because of imbalances in energy balance favouring energy intake. Whilst over 50% of a person's energy requirement goes towards the maintenance of physiological functions, around 40% is used for physical activity. In addition to this, around 10-15% of energy is spent on what is termed as Diet Induced Thermogenesis (DIT). Diet Induced Thermogenesis is the increase in energy expenditure following a meal, and represents the energy utilised for the digestion and metabolism of food. Some nutrients such as proteins require more energy to digest and therefore produce a greater DIT than others. In addition to this, some food components are able to independently stimulate calorie burning. For example caffeine, chilli, ginger and green tea have been shown to induce calorie burning through DIT. Therefore the inclusion of such foods in the diet could increase energy expenditure and thereby help in weight control.

The objective of this study is to determine the DIT effects of some plant foods that are native to Scotland (blackberries, blueberries, red raspberries, wild garlic and sea buckthorn). These foods have been shown to contain compounds that stimulate DIT. If found to be effective, these foods could then be used to develop dietary strategies for weight control in Scotland.

DETAILED DESCRIPTION:
Obesity prevalence is increasing around the world and the United Kingdom is no exception. Latest statistics show that approximately 25% of the UK population is obese and is predicted to rise to 70% by 2020 if present trends continue. Obesity is particularly widespread in Scotland where approximately 62% of the population are of a BMI over 25kg/m2. Curtailing obesity rates is a public health priority as excess weight is also the greatest predictor of other co-morbidities such as cardiovascular disease, cancer and diabetes, and hence collectively exerts a significant toll on the health and economic burden of the country.

Weight gain occurs primarily due to an imbalance in energy balance status where energy intake outweighs expenditure. Energy expenditure (EE) in adults consists of three components: basal metabolism (50-70% of EE), physical activity (30-40% of EE) and diet induced thermogenesis (DIT). The latter is described as the thermic effect of food and is the increase in EE above Basal Metabolic Rate after a meal, and usually ranges between 3-10% of total EE (depending on the composition of the meal). Whilst cornerstone approaches to weight control have focused on strategies to reduce energy intake and increase physical activity, the still escalating obesity levels show that this approach is ineffective in the long term possibly due to poor long-term compliance to dietary regimes and adequate physical activity. Thus it is being increasingly recognised that the most sustainable long-term strategy for reducing obesity is making small diet and lifestyle changes that would positively influence energy regulatory mechanisms targeted at preventing a positive energy balance. It is also now recognised that genetic predispositions to a slow mechanism characterised by a slow metabolic rate and capacity for fat oxidation also determines an individual's propensity to weight gain. Furthermore, studies have shown that weight loss and reduced food intake result in an attenuation of EE possibly due to the loss of lean mass and improved metabolic efficiency. The regular consumption of high DIT foods which could increase EE and fat oxidation whilst circumventing these energy sparing mechanisms may have significant potential in long-term weight control. Indeed studies demonstrating pronounced obesity in mice whose DIT mechanism were inactivated indicates the important role thermogenesis plays in weight control

Food components such as chilli (capsaicin), ginger, mustard, pepper, caffeine, green tea (flavanols) and medium-chain triglycerides have been demonstrated as increasing DIT. The thermogenic effects of these compounds have been shown to be mainly via the sympathetic nervous system. Pharmacological agents such as ephedrine and salicylate as well as food constituents such as methylxanthines (theophylline and caffeine) and caffeine have been shown to possess sympathomimetic properties and induce fat oxidation and thermogenesis in effector cells by stimulating the release of noradrenalin. Flavanoids such as green tea catechins have also been shown to stimulate this pathway. Sympathetically released noradrenalin has been shown to activate Beta3adrenoceptors and thereby induce thermogenesis and fat oxidation in peripheral tissues as well as activate uncoupling protein (UCP1) that mediates thermogenesis in brown adipose tissue (BAT). Plant phenolics have also been shown to demonstrate thermogenic effects, particularly Oleuropein, green tea catechins, Kaempferol, flavanol glycosides, stilbenes and quercetin.

The objective of the present pilot study is to assess the thermogenic effects of some plant foods native to Scotland that contain the above phytochemicals. Specifically, the study will investigate the thermogenic effects of berries (blackberries [Rubus sp.], blueberries [Vaccinium corymbosum] and red raspberries [Rubus idaeus L]), wild garlic (Allium ursinum) and sea buckthorn (Hippophae rhamnoides). Blackberries, blueberries and raspberries have been shown to be rich in flavonoids and phenolics including catechins and raspberry ketones which have been suggested to be thermogenic. These berries are also rich in anthocyanins such as cyanidin-3-glucoside which has been shown to potentially promote thermogenesis by upregulating UCP1. Furthermore, blueberries have been shown to be a good source of stilbenes such as resveratrol and pterostilbene which have demonstrated thermic effects elsewhere. Similarly, sea buckthorn has been reported to contain catechins, epicatechins and flavonols such as isorhamnetin, quercetin and kaempferol. Sea buckthorn is also rich in carotenoids, especially those with provitamin A activity that have been shown to upregulate the expression of UCP1 and thereby influence thermogenesis. Wild garlic contains Sulphur containing compounds such as alliin and Allicin derivatives (diallyldisulphide) that in studies using garlic have shown thermogenic activity by enhancing noradrenalin secretion and stimulating brown adipose tissue. Indeed the total thiosulfinate content in wild garlic has been shown to be comparable to garlic.

The presence of thermogenic compounds in these plant products logically suggests that they may have a thermic effect in humans and this forms the rationale for the present study. No studies have investigated the thermic effects of these foods in humans and their therapeutic potential in weight control from a thermogenesis perspective. The proposed pilot study will provide preliminary data on the thermic effects of these Scottish foods and provide a basis for future research.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged between 18-50 years
* Body mass index between 18.5 - 25.0 kg/m2

Exclusion Criteria:

* Suffering from thyroid disorders, metabolic/genetic diseases
* On prescription medications known to affect metabolism including hormonal contraceptives and thyroid medications
* Post-menopausal
* Allergic/intolerant to any foods
* Eating disorders
* Alcohol and/or other substance misuse issues
* Extreme intake of caffeine (more than 6 cups of tea and/or coffee per day)
* Smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Diet Induced Thermogenesis | Baseline then for 15 minutes hourly for 5 hours post prandial
  Measured as the difference in Resting Metabolic Rate (RMR) during fasting and postprandial states

SECONDARY OUTCOMES:
Substrate utilisation for energy metabolism | Baseline and hourly for 5 hours post prandial
  Based on the Respiratory Quotient (RQ) from RMR measurement and urinary urea, the proportion of carbohydrate, fat and protein used for energy production will be estimated.
Satiety and palatability of the test meals. | Immediately before and after consumption of the test meal.
  Measured using 100mm continuous-line scales anchored at each end with opposing answers to satiety and palatability related questions

CONTACTS AND LOCATIONS:
Overall Officials: Viren Ranawana, MSc, PhD, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen, Foresterhill, Aberdeen, AB25 2ZD, United Kingdom
Locations (1):
- Rowett Institute of Nutrition and Health, Human Nutrition Unit, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No